CLINICAL TRIAL: NCT05907122
Title: A Randomized, Double-blind Study Evaluating Pharmacokinetic Similarity of ABP 206 Compared With OPDIVO® (Nivolumab) in Resected Stage III or Stage IV Melanoma Subjects in the Adjuvant Setting
Brief Title: A Study to Evaluate Similarity of ABP 206 Compared With OPDIVO® (Nivolumab) in Subjects With Resected Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20220083
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Melanoma
Keywords: Pharmacokinetic similarity study; Adjuvant melanoma treatment; Advanced Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study is double-blinded; therefore, the investigators, study personnel (with the exception of the data monitoring committee, authorized unblinded sponsor and contract research organization staff, and unblinded site pharmacy staff), and the study subjects will remain blinded to treatment allocation. ABP 206 and nivolumab will be coded and labeled to protect blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ABP 206 (Experimental): Subjects will receive Dose A of ABP 206 via intravenous (IV) infusion.
  Interventions: Drug: ABP 206
- FDA-licensed Nivolumab (Active Comparator): Subjects will receive Dose A of FDA-licensed Nivolumab via IV infusion.
  Interventions: Drug: FDA-licensed Nivolumab
- EU-authorized Nivolumab (Active Comparator): Subjects will receive Dose A of EU-authorized Nivolumab via IV infusion.
  Interventions: Drug: EU-authorized Nivolumab

INTERVENTIONS:
Drug: ABP 206 — ABP 206 will be given intravenously over a period of 30 minutes, every 4 weeks (Q4W) for a total of 12 months.
  Arms: ABP 206
Drug: FDA-licensed Nivolumab — FDA-licensed Nivolumab will be given intravenously over a period of 30 minutes, Q4W for a total of 12 months.
  Other Names: OPDIVO®
  Arms: FDA-licensed Nivolumab
Drug: EU-authorized Nivolumab — FDA-licensed Nivolumab will be given intravenously over a period of 30 minutes, Q4W for a total of 12 months.
  Other Names: OPDIVO®
  Arms: EU-authorized Nivolumab

SUMMARY:
The purpose of this study is to investigate the pharmacokinetic (PK) similarity and efficacy, safety, and immunogenicity of ABP 206 compared with OPDIVO® (nivolumab) in subjects with resected advanced melanoma.

DETAILED DESCRIPTION:
Eligible subjects will be randomized in a 1:1:1 ratio to receive either ABP 206, Food and Drug Administration (FDA)-licensed nivolumab, or European Union (EU)-authorized nivolumab.

The treatment period is in alignment with the maximum treatment duration for OPDIVO® (nivolumab, reference product) in the adjuvant setting for melanoma.

All subjects will be treated until recurrence of disease, unacceptable toxicity, or subject withdrawal of consent with a maximum of 1 year of treatment.

The total duration of study participation for each subject will be approximately 13 months.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Completely removed melanoma by surgery performed within 12 weeks of randomization
* Advanced Melanoma
* Tumor tissue from the resected site of the disease must be available for biomarker analyses in order to be randomized
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1

Exclusion Criteria:

* Previous anti-cancer treatment
* Known hypersensitivity to monoclonal antibodies or to any of the excipients of the study drug
* Ocular or uveal melanoma or history of carcinomatosis meningitis
* History of auto-immune disease
* Subject has medical conditions requiring systemic immunosuppression with either corticosteroids or other immunosuppressive medications within 14 days of the first dose of the investigational product

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Area Under the Serum Concentration-time Curve from Time Zero to 28 Days (AUC0-28d) | Day 1 (Postdose) through Day 28
  The PK similarity (AUC0-28d) of ABP 206 compared with nivolumab will be demonstrated in subjects with advanced melanoma in the adjuvant setting.
Area Under the Serum Concentration-time Curve Over the Dosing Interval at Steady State (AUCtau_SS) | Week 17 through Week 21
  The PK similarity (AUCtau_ss) of ABP 206 compared with nivolumab will be demonstrated in subjects with advanced melanoma in the adjuvant setting.

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration Following the First Dose (Cmax_dose 1) | Week 1 (Baseline) through Week 9, Week 17 to 29, Week 41, and Week 53 (End of Study)
  The comparison of PK (Cmax_dose 1) of ABP 206 with nivolumab will be determined in subjects with advanced melanoma in the adjuvant setting.
Maximum Observed Serum Concentration at Steady State (Cmax_ss) | Week 1 (Baseline) through Week 9, Week 17 to 29, Week 41, and Week 53 (End of Study)
  The comparison of PK (Cmax_ss) of ABP 206 with nivolumab will be determined in subjects with advanced melanoma in the adjuvant setting.
Serum Concentrations at Predose (Ctrough) | Week 1 (Baseline) through Week 9, Week 17 to 29, Week 41, and Week 53 (End of Study)
  The PK similarity (Ctrough) of ABP 206 compared with nivolumab determined in subjects with advanced melanoma in the adjuvant setting.
Number of Subjects With Treatment-Emergent Serious Adverse Events | Week 1 (First dose of study drug) through Week 53 (End of Study)
  The safety (treatment-emergent serious adverse events) of ABP 206 compared with nivolumab will be assessed in subjects with advanced melanoma in the adjuvant setting.
Number of Subjects With Treatment-Emergent Adverse Events | Week 1 (First dose of study drug) through Week 53 (End of Study)
  The safety (treatment-emergent adverse events) of ABP 206 compared with nivolumab will be assessed in subjects with advanced melanoma in the adjuvant setting.
Number of Subjects With Treatment-emergent Adverse Events-of-interest | Week 1 (First dose of study drug) through Week 53 (End of Study)
  The safety (treatment-emergent adverse events-of-interest) of ABP 206 compared with nivolumab will be assessed in subjects with advanced melanoma in adjuvant setting.
Number of Subjects With Anti-drug Antibodies (ADAs) | Predose on Week 1 (Baseline), Weeks 5, 9, 17, 21, 29, 41, and at Week 53 (End of Study)
  The immunogenicity of ABP 206 compared with nivolumab will be assessed in subjects with advanced melanoma in the adjuvant setting.
Recurrence-free Survival (RFS) | Randomization through 12 months (or until RFS criteria is met)
  The RFS is assessed to compare the efficacy of ABP 206 with nivolumab in subjects with advanced melanoma in the adjuvant setting. The RFS is defined as the time between the date of randomization and the date of first recurrence (local, regional, distant metastasis) or death (whatever the cause), or date of last visit/contact with disease assessments (for subjects who remain alive and whose disease has not recurred).
Time to reach Cmax following the first dose (Tmax_dose 1) | Week 1 (Baseline) through Week 9, Week 17 to 29, Week 41, and Week 53 (End of Study)
  The comparison of PK (Tmax_dose 1) of ABP 206 with nivolumab will be determined in subjects with advanced melanoma in the adjuvant setting.
Time to reach Cmax at steady state (Tmax_ss) | Week 1 (Baseline) through Week 9, Week 17 to 29, Week 41, and Week 53 (End of Study)
  The comparison of PK (Tmax_SS) of ABP 206 with nivolumab will be determined in subjects with advanced melanoma in the adjuvant setting.
Serum Concentrations (Ctrough) | At Week 5 (Pre-dose), and at Weeks 17 and 21 (Pre-dose)
  The comparison of PK (Ctrough) of ABP 206 with nivolumab will be determined in subjects with advanced melanoma in the adjuvant setting.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (76):
- United States (2):
  - Cancer and Blood Specialty clinic, Long Beach, California
  - St. Vincent Frontier Cancer Center - Oncology, Billings, Montana
- Centro De Investigaciones Medicas Mar Del Plata (CIMMDP) - Rheumatology, Mar Del Plata, Río Negro Province, Argentina
- Bosnia and Herzegovina (5):
  - Clinical Center University of Sarajevo - Clinic of Oncology, Sarajevo, Kanton Sarajevo
  - University Clinical Centre of the Republic of Srpska - Gastroenterology, Banja Luka, Republika Srpska
  - University Clinical Center Tuzla - Oncology, Hematology and Radio, Tuzla, Tuzlanski Kanton
  - Cantonal hospital Zenica - Oncology, Zenica, Zeničko-dobojski Kanton
  - University Clinical Hospital Mostar - Clinic for Lung Diseases, Mostar
- Brazil (9):
  - ATO Oncologia, Fortaleza, Ceará
  - Hospital Sao Rafael, Salvador, Estado de Bahia
  - Hospital Sirio Libanes - Brasilia, Brasília, Federal District
  - Instituto de Oncologia do Parana, Curitiba, Paraná
  - CTO Centro de Tratamento Oncológico, Belém, Pará
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - CEPON - Centro de Pesquisas Oncológicas, Florianópolis, Santa Catarina
  - Fundacao Pio XII - Hospital de Cancer de Barretos - Hospital de Amor, Barretos, São Paulo
  - Faculdade de Medicina de Sao Jose do Rio Preto-SP (FAMERP) - Hospital de Base (HB) - Oncology, São Paulo
- Oncocentro APYS, Valparaíso, Región de Valparaíso, Chile
- Croatia (2):
  - KBC "Sestre milosrdnice", Grad Zagreb, City of Zagreb
  - University Hospital Centre Zagreb - Oncology department, Zagreb, City of Zagreb
- Georgia (2):
  - LTD "Israel-Georgian Medical Research Clinic Healthycore", Tbilisi
  - JSC "K.Eristavi National Center of Experimental and Clinical Surgery", Tbilisi
- Italy (4):
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori IRST S.R.L, Meldola, Forli
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Istituto Dermopatico dell'Immacolata (IDI) - IRCCS - Oncologia, Roma
  - Azienda ospedaliero Universitaria Senese - Policlinico Le Scotte, Siena
- Japan (8):
  - Nagoya City University Hospital - Dermatology, Nagoya, Aiti [Aichi]
  - Sapporo Medical University Hospital, Sapporo, Hokkaidô [Hokkaido]
  - National Hospital Organization Kagoshima Medical Center - Haematology, Kagoshima, Kagosima [Kagoshima]
  - Shizuoka Cancer Center - Dermatology, Kōtoku, Tôkyô [Tokyo]
  - Keio University Hospital - Dermatology, Shinjuku-ku, Tôkyô [Tokyo]
  - Kumamoto University Hospital - Dermatology, Kumamoto
  - Niigata Cancer Center Hospital - Dermatology, Niigata
  - Osaka International Cancer Institute - Dermatological Oncology, Osaka, Ôsaka [Osaka]
- National Cancer Institute - Conservative Tumour Therapy, Vilnius, Vilnius County, Lithuania
- Malaysia (6):
  - Hospital Pulau Pinang - Rheumatology, Pulau Pinang, Pahang
  - Hospital Umum Sarawak, Kuching, Sarawak
  - Institut Kanser Negara, Putrajaya, Selangor
  - Hospital Universiti Sains Malaysia, Kubang Kerian, Terengganu
  - Hospital Kuala Lumpur - Surgery, Kuala Lumpur, Wilayah Persekutuan Kuala Lump
  - Hospital Canselor Tuanku Muhriz UKM, Kuala Lumpur, Wilayah Persekutuan Kuala Lump
- Mexico (5):
  - Centro de Inm Onc de Occ Sa de Cv, Guadalajra, Jalisco
  - Althian - Research Management Center, San Pedro Garza García, Nuevo León
  - Hospital Angeles Centro Médico San Luis Potosí - Cardiologia, San Luis Potosí City, San Luis Potosí
  - ONCOCENTER PUEBLA - Dermatology, Puebla City
  - Clinical Research Institute, Tlalnepantla
- Arensia Exploratory Medicine - Moldova - IMSP Institutul Oncologic - Oncology, Chisinau, Moldova, Republic of, Moldova
- Amphia Hospital - unspecified, Breda, North Brabant, Netherlands
- Romania (2):
  - Arensia Exploratory Medicine - Romania - Institutul Oncologic Prof Dr Ion Chiricuta Cluj-Napoca - On, Cluj-Napoca, Cluj
  - Arensia Exploratory Medicine - Romania - Institutul Oncologic Prof Dr Alexandru Trestioreanu Bucures, Bucharest
- Serbia (3):
  - University Clinical Center of Nis, Clinic for Oncology, Niš, Nišavski Okrug
  - Institute for Oncology and Radiology of Serbia, Department for Lung Cancer, Belgrade
  - University Clinical Center of Kragujevac, Center for Internal Oncology, Kragujevac, Šumadijski Okrug
- South Africa (5):
  - The Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - Wits Clinical Research, Parktown, Johannesburg, Gauteng
  - Mary Potter Oncology Centre, Pretoria, Gauteng
  - Cape Gate Oncology Centre, Bellville, Western Cape
  - Cancercare - Rondebosch Oncology, Cape Town, Western Cape
- South Korea (5):
  - Inje University Haeundae Paik Hospital - Oncology, Busan, Busan Gwang'yeogsi [Pusan-Kwan
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggido [Kyonggi-do]
  - Severance Hospital, Yonsei University Health System - Division of Medical Oncology, Department of In, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
  - Asan Medical Center - Oncology, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
  - Samsung Medical Center - Family Medicine, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
- Spain (5):
  - Hospital San Pedro de Alcántara - Oncología, Cáceres, Cáceres
  - H.U.V.Arrixaca, El Palmar, Murcia, Región de
  - Hospital de la Santa Creu i Sant Pau - Oncología Médica, Barcelona
  - Hospital HLA Jerez Puerta Sur, Seville
  - Consorcio Hospital General Universitario de Valencia - Oncología, Valencia
- Taiwan (2):
  - China Medical University Hospital - Internal Medicine, Taichung, Taichung Municipality
  - Taipei Medical University - Shuang Ho Hospital Ministry of Health and Welfare, New Taipei City, Taipei
- Thailand (4):
  - Khon Kaen University, Srinagarind Hospital - Academic Clinical Research Office (ACRO), Khonkaen, Changwat Khon Kaen
  - Prince of Songkla University, Songkhla, Changwat Songkhla
  - King Chulalongkorn Memorial Hospital [Medical Oncology], Bangkok, Krung Thep Maha Nakhon [Bangko
  - Siriraj Hospital - Medical Oncology, Bangkok, Krung Thep Maha Nakhon [Bangko
- Vietnam (2):
  - Vietnam National Cancer Hopsital, Hanoi, Ha Noi, Thu Do
  - HCM Oncology Hospital - Medical Oncology, Ho Chi Minh City, Ho Chi Minh, Thanh Pho [Sai Go

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data-sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data-sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com